CLINICAL TRIAL: NCT05329701
Title: Individualized Duration of Antibiotic Treatment in Culture Negative Early Onset Infection in Term Born Newborns: A Nationwide Randomized Controlled Non-inferiority Trial.
Brief Title: Individualized Duration of Antibiotic Treatment in Early Onset Infection in Newborns.
Acronym: DurATi-n
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ulrikka Nygaard (Other)
Collaborators: Innovation Fund Denmark (Individual); University of Copenhagen (Other)
Responsible Party: Sponsor-Investigator, Ulrikka Nygaard, MD,Phd, Consultant, Associate Professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-21004823
Record Dates: First submitted 2022-04-07; First posted 2022-04-15 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Early-Onset Neonatal Sepsis; Antibiotic Side Effect
Keywords: neonatal; early-onset; infection; antibiotic
MeSH Terms: conditions — Neonatal Sepsis; Infections

STUDY DESIGN:
Intervention Model Description: The study is a nationwide multicenter open label non-inferiority pragmatic randomized controlled trial. Patients will be randomized 1:1 to experimental treatment duration or standard care. Patients will be stratified based on if maximum CRP level is above or below 90 mg/l.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Individualized treatment duration (Experimental): Antibiotic treatment will be discontinued when both of the following two criteria are fulfilled:
  1. The infant has had 24 hours without clinical symptoms of infection, after systematic clinical evaluation by a neonatologist. Clinical symptoms specified in Table 1.
  2. CRP is < 30 mg/l. If CRP is > 30 at the time when the infant has been symptom-free for 24 hours, CRP will be assessed once every 24 -48 hours and antibiotics will be stopped when CRP < 30.
  Interventions: Other: Individualized treatment duration strategy
- Standard treatment duration (No Intervention): Standard treatment duration is seven days.

INTERVENTIONS:
Other: Individualized treatment duration strategy — As listed under arm description.
  Arms: Individualized treatment duration

SUMMARY:
A nationwide multicenter open label randomized controlled non-inferiority trial, including 18 departments. The study aims to compare an individualized antibiotic treatment duration with standard seven days of antibiotic treatment for culture negative early-onset infection in term newborns.

DETAILED DESCRIPTION:
There is a documented antibiotic overuse in newborns, and a lack of evidence for the optimal duration of antibiotic therapy in culture-negative infection. The study aims to evaluate the effect of individualized treatment duration in early-onset infection.

The study aims to compare an individualized treatment duration with seven days of treatment for culture negative early-onset infection. The investigators hypothesize that the individualized treatment duration, based on structured clinical assessment of symptoms and level of CRP is non-inferior to the standard care being seven days of treatment. In the experimental treatment arm, antibiotics will be stopped when the participant had 24 hours without symptoms and at same time point have decreasing level of CRP, with an absolute threshold of CRP ≤ 30 mg/l. The investigators hypothesize that individualized treatment will shorten the duration of antibiotic therapy in newborns with early onset infection with very little risk of relapse. Newborns who fulfill criteria to stop antibiotics within 48 hours will not be eligible for inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age ≥ 35 weeks
* Birth weight ≥ 2000
* Probable or possible infection according to the structured infection risk assessment
* Sufficient size blood culture, preferably 0.5-1 ml, but at least 0.2 ml, drawn after onset of symptoms but before start of antibiotic treatment
* Negative blood culture after 48 hours

Exclusion Criteria:

* Infants with positive blood culture
* Blood culture volume prior to antibiotics of < 0.2 ml
* Site-specific infection as for example, meningitis or osteomyelitis
* Infant fulfill current recommendation to stop antibiotic treatment at 36-48 hours; Low suspicion of sepsis initially including few and vague symptoms, CRP maximum 35-50 mg/l, negative blood culture and no symptoms after 48 hours of treatment

Ages: 1 Hour to 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 488 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2025-04-05 (Actual); Study Completion 2025-08-10 (Actual)

PRIMARY OUTCOMES:
Readmission due to infection. | From 1-21 days after end of first course of antibiotic treatment.
  Readmission due to infection, defined as symptoms, affected biomarkers and antibiotic treatment > 72 hours
Death | From 1-21 days after end of first course of antibiotic treatment.
  Death of any cause
Total use of antibiotics | From initiation of antibiotics and the next 28 days.
  Use of antibiotics (in hours)

SECONDARY OUTCOMES:
C-reactive protein (CRP) | CRP measured at follow-up 2 days after initial antibiotic treatment ended
  CRP (mg/l) levels at follow-up
Readmission due to infection within 3 months | From 1-100 days after first course of antibiotics ended.
  Readmission due to infection, defined as symptoms, affected biomarkers and antibiotic treatment > 72 hours

OTHER OUTCOMES:
Hospital stay | From initiation of antibiotics and the next 28 days.
  Length of hospital stay within 28 days after initial antibiotic treatment started
Positive blood cultures | From 1-21 days after end of first course of antibiotic treatment.
  Numbers of culture positive infections
Serious adverse events (SAE) | From initiation of antibiotics and the next 100 days.
  Any serious adverse events related to the study intervention
Total use of antibiotics | From initiation of antibiotics and the next 100 days.
  Use of antibiotics (in hours)
Breastfeeding | At 2 day and 21 day follow up, after end of initial antibiotic treatment.
  Exclusive and partial breastfeeding rates

CONTACTS AND LOCATIONS:
Overall Officials: Emma Malchau Carlsen, MD, PhD, Principal Investigator — Department of Neonatology, Rigshospitalet, Copenhagen, Denmark; Tine Brink Henriksen, MD, Prof, Study Director — Department of Neonatology, Skejby Sygehus, Aarhus, Denmark
Locations (1):
- Ulrikka Nygaard, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Researchers who provide a methodologically sound proposal will be granted access to a full copy of individual deidentified data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available from 3 months after the publication of the study, ending 5 years after publication.
Access Criteria: Proposals should be directed to the corresponding author of this article, and access can be granted after the proposal is approved by the trial steering committee. Data will be available at a third party website after a data access agreement is signed (link to website will be shared after request is approved).

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-01-17): https://cdn.clinicaltrials.gov/large-docs/01/NCT05329701/SAP_000.pdf